CLINICAL TRIAL: NCT06882850
Title: Immunomodulation During Pregnancy Through Low-Dose Aspirin: a Hypothetical Mechanism for the Prevention of Preeclampsia?
Brief Title: Immunomodulation During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Ana Luisa Areia, Clinical Professor, Unidade Local de Saúde de Coimbra, EPE
Other Study IDs: OBS.SF.160/2022
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Aspirin; Pregnancy Complications; Immunology
Keywords: Immunology; Pregnancy; Aspirin; Lymphocytes; T-Lymphocytes
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy pregnancies: High-risk preeclampsia pregnencies

SUMMARY:
The goal of this observational study is to learn about the effects of low dose aspirin in immunity Pregnant women taking aspirin for other reasons (preeclampsia prevention) will be studied. The main question it aims to answer is: evaluate the effect of LDA on the modulation of innate immunity cells (NK cells, monocytes, γδ T cells) and/or acquired immunity (B and T lymphocytes, Treg cells, Th cells).

Participants already taking intervention A as part of their regular medical care for RA will answer online survey questions about their joint pain for 5 years.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effect of LDA on the modulation of innate immunity cells (NK cells, monocytes, γδ T cells) and/or acquired immunity (B and T lymphocytes, Treg cells, Th cells). The secondary objectives are to quantify pro-inflammatory and anti-inflammatory cytokines before and after LDA administration, as well as to assess maternal and fetal outcomes, comparing these parameters with those of low-risk PE pregnancies that do not require prophylactic LDA administration.

A prospective longitudinal study will be conducted, lasting a minimum of 40 weeks and a maximum of 24 months. Singleton pregnancies monitored at the Centro Hospitalar e Universitário de Coimbra will be included, with the first consultation occurring before 14 weeks of gestation and gestational age determined by first-trimester ultrasound. The study group will consist of women at high risk of PE according to clinical/historical criteria, who have not yet started LDA intake at the time of recruitment. Pregnant women will be classified as having a low or high risk of PE (risk of ≥ 1 in 50 for preterm PE) using the Fetal Medicine Foundation algorithm. This algorithm evaluates maternal clinical risk factors, mean arterial pressure (MAP), uterine artery pulsatility index (UtA-PI), and pregnancy-associated plasma protein A (PAPP-A). Women classified as high-risk will receive prophylactic aspirin (150 mg once daily).

As this is a preliminary study, 30 pregnant women will initially be included: 15 at high risk of PE (study group) and 15 at low risk (control group). Peripheral blood samples will be collected from both groups, utilizing routine pregnancy blood draws, at three time points (1st, 2nd, and 3rd trimesters). This will allow the evaluation of fluctuations in immune cells (NK cells, B and T lymphocytes, Treg cells, Th cells) and cytokine levels (IL-1, IL-6, IL-8, TNF-α, INF-γ, TGF-β, and IL-10). In high-risk PE pregnancies, additional peripheral blood samples will be collected before LDA administration and four weeks afterward.

Flow cytometry methodology will be used to determine immune cell frequencies, while plasma cytokine levels will be measured using ELISA and Luminex methodologies. After delivery, in both groups, histopathological evaluation (immunohistochemical staining) of the placenta will be performed, analyzing the aforementioned immune cells, as well as umbilical cord blood analysis using flow cytometry.

ELIGIBILITY:
Inclusion Criteria: - Singleton pregnancy

* Patients attending prenatal consultations at the Obstetrics Service A of CHUC, with the first consultation occurring before 14 weeks of gestation
* Gestational age determined by first-trimester ultrasound
* Study group: Women classified as high risk for PE according to clinical/historical criteria and the Fetal Medicine Foundation algorithm. LDA-naïve.

Exclusion Criteria: Multiple pregnancy

* Autoimmune diseases
* Prior use of LDA or other immunomodulatory medication before potential recruitment
* History of spontaneous miscarriages and/or medical termination of pregnancy
* Fetal malformation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant female
Study Population: Women attending routine low-risk prenatal consultations at the Department of Obstetrics of the Centro Hospitalar Universitário de Coimbra (CHUC).
  A written procedure detailing the research and the general objectives of the proposal will be submitted to the hospital's ethics committee for approval. Informed consent from patients will be obtained under strict ethical protocols.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of Low dose aspirin (LDA) on the modulation of immunity cells | 30 weeks
  innate immunity cells and/or acquired immunity
Th1, Th2, Treg, Th17, and Th1/17 | 30 weeks
  Absolute and relative frequencies in total lymphocytes (LY, x10⁹/L; %)

SECONDARY OUTCOMES:
Maternal outcomes | 30 weeks
  Maternal Complications: Gestational diabetes, gestational hypertension, preterm birth
Maternal outcomes | 30 weeks
  Weeks of Delivery
Maternal outcomes | 30 weeks
  Type of delivery (vaginal or cesarean section)

OTHER OUTCOMES:
Fetal Complications | 30 weeks
  Preterm birth Neonatal intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Ana L Areia, PhD MD, Principal Investigator — University of Coimbra
Locations (1):
- Unidade Local de Saúde de Coimbra, E.P.E., Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All of my research in the form of an article with the whole protocol and results
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From My 2025 to May 2030

REFERENCES:
- [Background] 1. Cadavid AP. Aspirin: The Mechanism of Action Revisited in the Context of Pregnancy Complications. Front Immunol. 2017;8:261. 2. Mittelberger J, Seefried M, Franitza M, Garrido F, Ditsch N, Jeschke U, et al. The Role of the Immune Checkpoint Molecules PD-1/PD-L1 and TIM-3/Gal-9 in the Pathogenesis of Preeclampsia-A Narrative Review. Medicina (Kaunas). 2022;58(2). 3. Khanabdali R, Shakouri-Motlagh A, Wilkinson S, Murthi P, Georgiou HM, Brennecke SP, et al. Low-dose aspirin treatment enhances the adhesion of preeclamptic decidual mesenchymal stem/stromal cells and reduces their production of pro-inflammatory cytokines. J Mol Med (Berl). 2018;96(11):1215-1225. 4. Panagodage S, Yong HE, Da Silva Costa F, Borg AJ, Kalionis B, Brennecke SP, et al. Low-Dose Acetylsalicylic Acid Treatment Modulates the Production of Cytokines and Improves Trophoblast Function in an in Vitro Model of Early-Onset Preeclampsia. Am J Pathol. 2016;186(12):3217-3224. 5. Robillard PY, Dekker G, Scioscia M, Saito S. Progress in the understanding of the pathophysiology of immunologic maladaptation related to early-onset preeclampsia and metabolic syndrome related to late-onset preeclampsia. Am J Obstet Gynecol. 2022;226(2S):S867-S875. 6. Brox R, Hackstein H. Physiologically relevant aspirin concentrations trigger immunostimulatory cytokine production by human leukocytes. PLoS One. 2021;16(8):e0254606. 7. Dong W, Yin L. Expression of lipoxin A4, TNFalpha and IL-1beta in maternal peripheral blood, umbilical cord blood and placenta, and their significance in pre-eclampsia. Hypertens Pregnancy. 2014;33(4):449-456. 8. Tung YT, Wei CH, Yen CC, Lee PY, Ware LB, Huang HE, et al. Aspirin Attenuates Hyperoxia-Induced Acute Respiratory Distress Syndrome (ARDS) by Suppressing Pulmonary Inflammation via the NF-kappaB Signaling Pathway. Front Pharmacol. 2021;12:793107. 9. Dong W, Liu X, Liu W, Wang C, Zhao S, Wen S, et al. Dual antiplatelet therapy improves functional recovery and inhibits inflammation after ce
- [Derived] Areia AL, Almeida J, Alves V, Mota-Pinto A, Sa H. Modulation of Immune Cells by Aspirin During Pregnancy. Immunology. 2026 Feb;177(2):329-338. doi: 10.1111/imm.70051. Epub 2025 Oct 14. PMID 41087834